CLINICAL TRIAL: NCT04389294
Title: Hospital for Special Surgery COVID-19 Antibody Serology Among Anesthesiologists and Surgeons 2020
Brief Title: HSS Covid-19 Antibody Serology Among Surgeons & Anesthesiologists
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital for Special Surgery, New York (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 2020-0850
Record Dates: First submitted 2020-05-08; First posted 2020-05-15 (Actual); Results first posted 2024-01-03 (Actual); Last update posted 2024-01-03 (Actual); Status verified 2023-03

CONDITIONS: COVID

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: SARS-CoV2 serum antibody testing — Participants will have SARS-CoV2 serum antibody testing performed twice within 4 months of each other.

SUMMARY:
The goal of this study is to understand the infectious exposure of SARS-coronavirus 2 (SARS-CoV2) among surgeons and anesthesiologists and to correlate this status with self-reported indices of COVID-19 illness.

ELIGIBILITY:
Inclusion Criteria:

* Accredited to practice at HSS
* All anesthesiology and surgery faculty
* All anesthesia and orthopedic surgery fellows
* All orthopedic surgery residents

Exclusion Criteria:

• Refusal to participate in either of the interventions at either of the timepoints of interest

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 143 (Actual)
Dates: Start 2020-05-05 (Actual); Primary Completion 2020-06-16 (Actual); Study Completion 2020-09-04 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital for Special Surgery, New York, New York, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Surgeons and Anesthesiologists: Surgeons and anesthesiologists at a specialty orthopaedic hospital
Period: Overall Study
Arm/Group | Surgeons and Anesthesiologists
Started | 143
Completed | 143
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: All attending surgeons, anesthesiologists, and trainees in both departments (orthopedic surgery fellows, anesthesiology fellows and orthopedic surgery residents) as identified via an institutional listserv.
Arm/Group | Surgeons and Anesthesiologists
Number analyzed (Participants) | 143
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 125
  >=65 years | 18
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 41.4 [33 to 50.5]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 26
  Male | 117
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 28
  Not Hispanic or Latino | 109
  Unknown or Not Reported | 6
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2
  Asian | 20
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 8
  White | 110
  More than one race | 0
  Unknown or Not Reported | 3
Region of Enrollment [Number; unit: participants]
  United States | 143
Seroprevalence of SARS-CoV-2 IgG antibodies by serology testing [Count of Participants; unit: Participants] — The seroprevalence of severe acute respiratory syndrome coronavirus-2 (SARS-CoV-2) immunoglobulin G (IgG) antibodies among surgeons and anesthesiologists and associated antibody status with coronavirus disease 2019 (COVID-19) clinical illness was measured.
  Participants | 14

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With SARS-CoV-2 IgG Antibodies
Description: Prevalence of SARS-CoV-2 IgG antibodies by serology testing in participants at the time of study enrollment or 3 months later
Time Frame: Serology Test #1 (Study Enrollment) and Test #2 (3 months apart)
Population: Participating surgeons and anesthesiologists at a specialty orthopaedic hospital
Measure: Count of Participants; unit: Participants
Arm/Group | Surgeons and Anesthesiologists
Number analyzed (Participants) | 143
Participants | 14

2. Secondary Outcome: Differences in Sex Between IgG Antibody-positive vs. Negative Participants
Description: Secondary outcomes included differences in the survey responses between IgG antibody-positive and -negative participants. These included demographics such as sex.
Time Frame: Survey completed before or on day of serology testing asking about information from January 1, 2020 to May 5, 2020
Population: All surgeon and anesthesiologist participants with complete survey and serology testing data
Measure: Count of Participants; unit: Participants
Arm/Group | Surgeons and Anesthesiologists
Number analyzed (Participants) | 143
Participants
  SARS-CoV-2 IgG Positive Females | 2
  SARS-CoV-2 IgG Negative Females | 24
  SARS-CoV-2 IgG Positive Males | 12
  SARS-CoV-2 IgG Negative Males | 105

3. Secondary Outcome: Number of Asymptomatic Participants With Positive Antibody Serology
Description: Number of asymptomatic participants with positive antibody serology at either the study enrollment timepoint or 3 month timepoint
Time Frame: Serology Test #1 (Study Enrollment) and Serology Test #2 (3 months apart)
Population: Number of asymptomatic participants with positive antibody serology (n=89/143)
Measure: Count of Participants; unit: Participants
Arm/Group | Surgeons and Anesthesiologists
Number analyzed (Participants) | 89
Participants | 2

4. Secondary Outcome: Percentage of Antibody-positive Participants Who Subsequently Develop COVID-19
Description: Percentage of antibody-positive participants who subsequently develop COVID-19 at either the study enrollment timepoint or the 3 months time point
Time Frame: Serology Test #1 (Study Enrollment) and Serology Test #2 (3 months apart)
Population: Symptomatic participants who were antibody-positive
Measure: Count of Participants; unit: Participants
Arm/Group | Surgeons and Anesthesiologists
Number analyzed (Participants) | 54
Participants | 12

5. Secondary Outcome: Differences in Race Between IgG Antibody-positive vs. Negative Participants
Description: Secondary outcomes included differences in the survey responses between IgG antibody-positive and -negative participants. These included demographics such as race.
Time Frame: Survey completed before or on day of serology testing asking about information from January 1, 2020 to May 5, 2020
Population: All surgeon and anesthesiologist participants with complete survey and serology testing data
Measure: Count of Participants; unit: Participants
Arm/Group | Surgeons and Anesthesiologists
Number analyzed (Participants) | 143
Participants
  SARS-CoV-2 IgG Positive Whites | 10
  SARS-CoV-2 IgG Negative Whites | 99
  SARS-CoV-2 IgG Positive Blacks or African Americans | 2
  SARS-CoV-2 IgG Negative Blacks or African Americans | 6
  SARS-CoV-2 IgG Positive Asians | 2
  SARS-CoV-2 IgG Negative Asians | 18
  SARS-CoV-2 IgG Positive Others/Unknown | 0
  SARS-CoV-2 IgG Negative Others/Unknown | 6

6. Secondary Outcome: Differences in Average Number of Adults in Household Between IgG Antibody-positive vs. Negative Participants
Description: Secondary outcomes included differences in the survey responses between IgG antibody-positive and -negative participants. These included demographics such as number of adult household members.
Time Frame: Survey completed before or on day of serology testing asking about information from January 1, 2020 to May 5, 2020
Population: All surgeon and anesthesiologist participants with complete survey and serology testing data
Measure: Count of Participants; unit: Participants
Arm/Group | Surgeons and Anesthesiologists
Number analyzed (Participants) | 143
Participants
  SARS-CoV-2 IgG Positive | 14
  SARS-CoV-2 IgG Negative | 129

7. Secondary Outcome: Differences in Comorbidities Between IgG Antibody-positive vs. Negative Participants
Description: Secondary outcomes included differences in the survey responses between IgG antibody-positive and -negative participants. These included comorbidities.
Time Frame: Survey completed before or on day of serology testing asking about information from January 1, 2020 to May 5, 2020
Population: All surgeon and anesthesiologist participants with complete survey and serology testing data
Measure: Count of Participants; unit: Participants
Arm/Group | Surgeons and Anesthesiologists
Number analyzed (Participants) | 143
Participants
  SARS-CoV-2 IgG Positive Hypertension | 0
  SARS-CoV-2 IgG Negative Hypertension | 13
  SARS-CoV-2 IgG Positive Diabetes Mellitus | 0
  SARS-CoV-2 IgG Negative Diabetes Mellitus | 1
  SARS-CoV-2 IgG Positive Pulmonary Disease | 1
  SARS-CoV-2 IgG Negative Pulmonary Disease | 9
  SARS-CoV-2 IgG Positive CAD/Cardiac Condition | 0
  SARS-CoV-2 IgG Negative CAD/Cardiac Condition | 3
  SARS-CoV-2 IgG Positive Immunocompromised | 0
  SARS-CoV-2 IgG Negative Immunocompromised | 3
  SARS-CoV-2 IgG No Listed Comorbidities | 113

8. Other Pre Specified Outcome: Participants Who Were Eligible for in Plasma Donation
Description: Individuals who tested positive for COVID-19 who may be eligible for convalescent plasma donation
Time Frame: Serology Test #1 (Study Enrollment) and Test #2 (3 months apart)
Population: Surgeons and anesthesiologists who completed both the survey and serology testing
Measure: Count of Participants; unit: Participants
Arm/Group | Surgeons and Anesthesiologists
Number analyzed (Participants) | 143
Participants | 14

ADVERSE EVENTS:
Time Frame: Adverse event data was not collected
Description: Adverse event data was not collected
Arm/Group | Surgeons and Anesthesiologists
All-Cause Mortality (participants affected / at risk) | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-10-15): https://cdn.clinicaltrials.gov/large-docs/94/NCT04389294/Prot_SAP_000.pdf